CLINICAL TRIAL: NCT05630235
Title: Effects of a Hemp-derived Cannabidiol and Cannabidiolic-acid Oral Extract on Resting-state Electroencephalography and Neuropathic Pain Symptoms in People With Spinal Cord Injury
Brief Title: Effects of CBD/CBD-A Oral Extract on Resting-state EEG and Neuropathic Pain Symptoms After SCI
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Consortium for Medical Marijuana Clinical Outcomes Research (Other)
Responsible Party: Principal Investigator, Eva Widerstrom-Noga, Research Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20220782
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: SCI - Spinal Cord Injury; Neuropathic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBD/CBD-A followed by placebo group (Experimental): Participants in this group will receive a one time dose of CBD/CBD-A on visit 2, followed by a placebo on visit 3 after a two-week period.
  Interventions: Drug: CBD/CBD-A; Other: Placebo
- Placebo followed by CBD/CBD-A group (Experimental): Participants in this group will receive a placebo on visit 2, followed by a one time of CBD/CBD-A on visit 3 after a two-week period.
  Interventions: Drug: CBD/CBD-A; Other: Placebo

INTERVENTIONS:
Drug: CBD/CBD-A — Participants will be administered a one-time dose of 204.6 mg of CBD/CBD-A orally.
Other: Placebo — The placebo equivalent of the CBD/CBD-A dose administered orally.

SUMMARY:
The main purposes of this study are to (1) measure the effect of CBD/CBD-A on pain symptoms, pain intensity, pain unpleasantness, and skin sensitivity to hot and cold temperatures; and (2) measure the effect of CBD on brain electrical activity with electroencephalography (EEG).

ELIGIBILITY:
Inclusion Criteria:

1. Men or Women;
2. 18-64 years of age with an incomplete or complete acquired traumatic SCI;
3. Must have experienced neuropathic pain for a minimum of three months before entering the study (neuropathic pain will be assessed using the International SCI Pain Classification);
4. The pain intensity must be in the moderate to severe category, which will be defined as a score of at least four on an NRS (range of 0 to 10).
5. Must have previous experience with consuming cannabis and or cannabinoids.

Exclusion Criteria:

1. Current drug (DAST-10: >6) or alcohol abuse (AUDIT: >10);
2. Current use of cannabis plant or cannabis products (CBD or CBD+THC) or any other drugs of abuse (unless prescribed) including alcohol;
3. Presence of significant medical illness (e.g., diabetes, obesity, cardiovascular disease, hypertension, hepatitis) or other significant neurological trauma;
4. History of or current severe psychopathology (e.g., major depressive disorder, bipolar disorder, schizophrenia, post-traumatic stress disorder) judged by the investigator to put the subject at greater risk of experiencing an adverse event;
5. Adults who are unable to consent, women who are pregnant, breastfeeding, or not practicing an effective form of birth control (condoms, diaphragm, birth control pill, IUD), and prisoners;
6. Current pregnancy. Pregnancy will be evaluated using a pregnancy test during the first study visit. Female subjects of childbearing potential will be required to use two forms of effective birth control for the 3 months prior to participating in the study and continuing for 1 month after completion of the study;
7. Have a history of renal or hepatic disease: or
8. Have elevated serum creatinine above the laboratory upper limit of normal (ULN): or
9. Have elevated serum transaminases (ALT or AST) above the ULN: or
10. Have elevated total bilirubin above the ULN; or
11. Take valproate, due increased risk of liver enzyme elevation; or
12. Currently using strong CYP2C19 and CYP3A4 inducers; or
13. Have suicidal ideation (subjects should be screened for suicidal ideation); or
14. Cannot abstain from the use of alcohol during the study period, due to increased risk of sedation; or
15. Have a known or suspected hypersensitivity to cannabidiol or tetrahydrocannabinol.
16. Have a known or suspected hypersensitivity to sesame seed oil, lecithin, or bovine gelatin.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in neuropathic pain intensity or unpleasantness. | Baseline, approximately 3 hours post intervention, and approximately 6 hours post intervention
  Assess changes in pain intensity and unpleasantness of the worst neuropathic pain using a numerical rating scale from 0-10 (0 no pain and 10 worst imaginable/unpleasant pain).
Change in brain electrocortical activity at rest. | Baseline and 3 hours post intervention
  Assess brain electrocortical activity at rest using a 64-channel Biosemi EEG system and conducting EEG power spectrum analysis

SECONDARY OUTCOMES:
Change in neuropathic pain symptoms severity using the NPSI. | Baseline, approximately 3 hours post intervention, and approximately 6 hours post intervention
  The Neuropathic Pain Symptom Inventory (NPSI) will assess the presence and severity of common neuropathic pain symptoms. Range 0-100 with higher scores representing greater neuropathic pain symptoms.
Change in sensory function using QST. | Baseline and 3 hours post intervention
  Sensory function will be assessed using quantitative sensory testing (QST) using an FDA-approved Thermal Sensory Analyzer.
Change in state anxiety using the STAI. | Baseline, approximately 3 hours post intervention, and approximately 6 hours post intervention
  Using the State-trait Anxiety Inventory (STAI), we will evaluate changes in momentary anxiety with scores ranging from 5-20. Higher values equate to greater anxiety symptoms.
Subjective Drug Effects | Baseline, approximately 3 hours post intervention, and approximately 6 hours post intervention
  Drug Effects Questionnaire (DEQ): The DEQ is a brief five item instrument used to assess subjective drug effects. The five items are presented on a 100 mm visual analogue scale ranging from not at all to extremely. The participants are instructed to draw a vertical line at any place between the two responses

CONTACTS AND LOCATIONS:
Overall Officials: Eva Widerstrom-Noga, PhD, DDS, Principal Investigator — University of Miami
Locations (1):
- Lynn Rehabilitation Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No